CLINICAL TRIAL: NCT04664205
Title: Metabolic, Hormonal, and Physiological Characterization of Isoenergetic High Intensity Interval Training and Moderate Intensity Continuous Training in Adults With Type I Diabetes
Brief Title: Isoenergetic High Intensity Interval Training and Moderate Intensity Training in Adults With Type I Diabetes
Acronym: HI1T
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: North Carolina Diabetes Research Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 20-3100
Record Dates: First submitted 2020-12-04; First posted 2020-12-11 (Actual); Results first posted 2024-07-26 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2022-02

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — High-Intensity Interval Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High intensity interval training, Moderate Intensity Continuous Training, Control (Experimental): Participants randomly assigned to this arm will first receive high intensity interval training and then randomly assigned to both moderate intensity continuous training and control session, on different days.
  Interventions: Other: High Intensity Interval Exercise; Other: Moderate Intensity Continuous Exercise; Other: Control
- Moderate Intensity Continuous Training, High Intensity Training, Control (Experimental): Participants randomly assigned to this arm will first receive moderate intensity continuous training then randomly assigned to both high intensity interval training and a control session, on different days.
  Interventions: Other: High Intensity Interval Exercise; Other: Moderate Intensity Continuous Exercise; Other: Control
- Control session, High intensity interval training, moderate intensity continuous training (Experimental): Participants randomly assigned to this arm will first complete a control session (no exercise) and then randomly assigned to both by a high intensity interval training and moderate intensity continuous training session, on different days.
  Interventions: Other: High Intensity Interval Exercise; Other: Moderate Intensity Continuous Exercise; Other: Control

INTERVENTIONS:
Other: High Intensity Interval Exercise — One session of high intensity interval exercise
Other: Moderate Intensity Continuous Exercise — One session of calorically matched moderate intensity exercise
Other: Control — No exercise, resting measures

SUMMARY:
Type 1 diabetes (T1D) is associated with increased risk of poor cardiometabolic health. Regular exercise is recommended for optimal management of comorbidities in T1D. Unique barriers to exercise exist for T1D, including fear of hypoglycemia, unpredictable glycemic excursions with exercise, and inadequate knowledge about exercise. Unlike traditional moderate intensity continuous training (MICT) which requires extended periods of time, high intensity interval training (HIIT) requires minimal time (~10 minutes of exercise per session), with the potential to rapidly stimulate mitochondrial biogenesis and metabolism. The extent to which these exercise strategies alter metabolomic signatures of carbohydrate, fat, and amino acid metabolism in T1D is unknown. The overall goal of the proposed project is to identify the acute metabolic effects and physiological modifiers of HIIT compared to MICT and control (CON) using metabolomic profiling and cardiometabolic assessments in 14 adults with T1D. Using a randomized cross-over approach, the primary aim is to compare the metabolomics response immediately post, 1 hr post, and glycemic control through 48 hrs after HIIT, compared to MICT matched for total energy expenditure, versus a no exercise CON. An additional aim will be to characterize the influence of biological sex and physiological outcomes (i.e. body composition, lean mass, visceral fat) on the metabolomics profile of these subjects. Outcomes from the present study, with existing data from our team, will lay the foundation for a larger diet and exercise lifestyle intervention that will ultimately lead to changes in clinical practice to co-manage glycemia and cardiometabolic comorbidities.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of presumed autoimmune T1D, receiving daily insulin
* Last hemoglobin A1c <9%
* 18-51 years
* Duration of T1D: ≥ 1 year
* Body mass index (BMI) <30 kg/m^2
* Generally healthy, with no conditions that could influence the outcome of the trial, and in the judgement of the investigators is a good candidate for the study, based on a review of health history

Exclusion Criteria:

* Physician diagnosis of active diabetic retinopathy that could be worsened by exercise
* Physician diagnosis of peripheral neuropathy with insensate feet
* Physician diagnosis of autonomic neuropathy
* Medications: beta-blockers, agents that affect hepatic glucose production such as beta adrenergic agonists, xanthine derivatives; any hypoglycemic agent other than insulin.
* Severe hypoglycemic event defined as the individual requiring a third party of hospitalization in the last 6 months
* Diabetic ketoacidosis in the last 6 months
* Has a closed-loop pump and not willing to use manual mode
* Physician diagnosis of cardiovascular disease that would affect exercise tolerance
* Currently doing HIIT
* Severely impaired hearing or speech
* Pregnancy

Ages: 18 Years to 51 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 14 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-09-15 (Actual); Study Completion 2022-09-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Abbie Smith-Ryan, PhD, Principal Investigator — University of North Carolina
Locations (1):
- Applied Physiology Laboratory, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 12 to 24 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Supporting Information: Study Protocol
Time Frame: Beginning 1 year and ending 2 years following article publication
Access Criteria: IRB, IEC, or REB approval, as applicable, and an executed data use/sharing agreement with UNC.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This was a cross-over design with all participants completing all treatments.
Period: First Exercise Session
Arm/Group | High Intensity Interval Training, Moderate Intensity Continuous Training, Control | Moderate Intensity Continuous Training, High Intensity Training, Control | Control Session, High Intensity Interval Training, Moderate Intensity Continuous Training
Started | 6 | 5 | 3
Completed | 6 | 5 | 3
Not Completed | 0 | 0 | 0
Period: Second Exercise Session
Arm/Group | High Intensity Interval Training, Moderate Intensity Continuous Training, Control | Moderate Intensity Continuous Training, High Intensity Training, Control | Control Session, High Intensity Interval Training, Moderate Intensity Continuous Training
Started | 6 | 5 | 3
Completed | 6 | 5 | 3
Not Completed | 0 | 0 | 0
Period: Third Exercise Session
Arm/Group | High Intensity Interval Training, Moderate Intensity Continuous Training, Control | Moderate Intensity Continuous Training, High Intensity Training, Control | Control Session, High Intensity Interval Training, Moderate Intensity Continuous Training
Started | 6 | 5 | 3
Completed | 6 | 5 | 3
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: All participants were randomly assigned to receive control session, high intensity interval training, and moderate intensity continuous training on different days.
  High Intensity Interval Exercise: One session of high intensity interval exercise
  Moderate Intensity Continuous Exercise: One session of calorically matched moderate intensity exercise
  Control: No exercise, resting measures
Arm/Group | All Participants
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 12
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 14
Percent Body Fat [Mean (Standard Deviation); unit: percent body fat] — Body fat percentage determined from whole body dual energy x-ray absorptiometry
  percent body fat | 26.6 (11.0)

OUTCOME MEASURES:

1. Primary Outcome: Mean Energy Expenditure Between HIIT and MICT
Description: Energy expenditure measured via indirect calorimetry (kcals) during exercise.
Time Frame: During exercise
Population: There was no exercise during the control session; therefore, this outcome does not apply for control trial.
Measure: Mean (Standard Deviation); unit: kcal
Groups:
- High Intensity Interval Training: High Intensity Interval Exercise: One session of high intensity interval exercise
- Moderate Intensity Continuous Training: Moderate Intensity Continuous Exercise: One session of calorically matched moderate intensity exercise
- Control Session: Control: No exercise, resting measures
Arm/Group | High Intensity Interval Training | Moderate Intensity Continuous Training | Control Session
Number analyzed (Participants) | 14 | 14 | 0
kcal | 264.5 (80.9) | 225.5 (57.4) |
Statistical Analysis 1: Comparison: High Intensity Interval Training vs Moderate Intensity Continuous Training; Test type: Superiority; p = 0.010, t-test, 2 sided

2. Primary Outcome: Difference in Mean Lactate During Exercise as an Indicator of Carbohydrate Metabolism
Description: Lactate measured using capillary finger prick (mmol/L).
Time Frame: Baseline, 1 hour post exercise
Population: There was no exercise during the control session; therefore, this outcome does not apply for control trial.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | High Intensity Interval Training | Moderate Intensity Continuous Training | Control Session
Number analyzed (Participants) | 14 | 14 | 0
mmol/L
  During exercise | 8.46 (2.83) | 7.11 (2.19) |
  1 hour post | 2.30 (1.05) | 1.75 (0.46) |
Statistical Analysis 1: Comparison: High Intensity Interval Training vs Moderate Intensity Continuous Training; Test type: Superiority; p = 0.069, ANCOVA

3. Secondary Outcome: Change in Continuous Glucose After Exercise Into Overnight
Description: Glucose monitoring using a continuous glucose monitor (mg/dL). Overnight values were collected based on the average mid-point of participants' sleep.
Time Frame: Immediately post-exercise and Overnight
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | High Intensity Interval Training | Moderate Intensity Continuous Training | Control Session
Number analyzed (Participants) | 14 | 14 | 14
mg/dL
  Immediately post exercise | 155.2 (11.3) | 146.9 (8.0) | 124.5 (6.3)
  Overnight | 139.7 (18.7) | 165.6 (6.0) | 150.3 (7.6)
Statistical Analysis 1: Comparison: High Intensity Interval Training vs Moderate Intensity Continuous Training vs Control Session; Test type: Superiority; p = 0.478, ANOVA

ADVERSE EVENTS:
Time Frame: From the time of signing the informed consent through the end of the study, a total of up to approximately 1 month
Arm/Group | High Intensity Interval Training | Moderate Intensity Continuous Training | Control Session
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/14 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 0/14 | 0/14 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-09-17): https://cdn.clinicaltrials.gov/large-docs/05/NCT04664205/Prot_SAP_000.pdf
  • Informed Consent Form (2021-09-17): https://cdn.clinicaltrials.gov/large-docs/05/NCT04664205/ICF_001.pdf